CLINICAL TRIAL: NCT04751617
Title: Impact of Pulmonary Rehabilitation on Quality of Life, Body Composition and Respiratory Function of Patients With a History of COVID-19
Brief Title: Pulmonary Rehabilitation of Patients With a History of COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Justyna Wyszyńska, Principal Investigator, University of Rzeszow
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rehabilitation after COVID-19
Record Dates: First submitted 2021-02-05; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Covid19
Keywords: SARS-CoV-2; Pulmonary rehabilitation; Quality of life; Body composition; Spirometry; Computed tomography; Morphology; Gasometry
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulmonary rehabilitation (intervention) (Experimental): This group will be covered by pulmonary rehabilitation.
  Interventions: Procedure: Pulmonary rehabilitation

INTERVENTIONS:
Procedure: Pulmonary rehabilitation — Pulmonary rehabilitation will include: early mobilization with frequent posture changes and simple exercises in bed taking into account the patient's respiratory tract. Respiratory physiotherapy will also include improving diaphragm function along with training additional respiratory muscles. Active exercises of the upper limbs will be accompanied by gradual muscle strengthening. Aerobic regeneration will be carried out by walking along the hospital corridor, stationary bike and climbing stairs. Body balance therapy in closed systems in front of the mirror will also be included. After kinesiotherapy, the session will end with a vibration massage and relaxation of the whole body. Motivational breathing training will be used every 2 hours, 7 days a week, performed independently by the patient in the ward room. The physiotherapy process will be carried out 6 times a week and lasts 30-45 minutes a day. The duration of rehabilitation depends on the patient's condition: from 7 to 14 days.

SUMMARY:
This study will determine the impact of pulmonary rehabilitation on quality of life, body composition and respiratory function in patients with a history of COVID-19.

DETAILED DESCRIPTION:
In December 2019, a novel coronavirus, SARS-CoV-2, appeared, causing a wide range of symptoms, mainly respiratory infection. In March 2020, the World Health Organization (WHO) declared Coronavirus Disease 2019 (COVID-19) a pandemic. COVID-19 has spread rapidly over several months, affecting patients across all age groups and geographic areas. The disease has a diverse course; patients may range from asymptomatic to those with respiratory failure, complicated by acute respiratory distress syndrome.

The main objective of this study is to assess the impact of pulmonary rehabilitation on quality of life, body composition and respiratory function in patients with a history of COVID-19.

The patients after COVID-19 will be included in the pulmonary rehabilitation protocol. The duration of rehabilitation will depend on the patient's condition: from 7 to 14 days.

Measurements:

* quality of life (WHOQoL-BREF)
* body composition (bioelectrical impedance analysis, BC-420 MA, Tanita)
* weight, height and BMI
* spirometry (Spirometr PNEUMO, abcMED)
* diffusion lung capacity for carbon monoxide (LUNGTEST 1000)
* morphology (CRP, D-Dimer, WBC) and gasometry (pCO2, pO2)
* chest computed tomography (CT).

These parameters will be recorded before the first day of rehabilitation (baseline), after completion of rehabilitation protocol, and three months after completion the rehabilitation protocol. A change in evaluated parameters will be assessed.

This will be a prospective, interventional, non-randomized study. All patients will be enrolled by Podkarpackie Center for Lung Diseases in Rzeszów.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients treated in Provincial Clinical Hospital No. 1 in Rzeszów/ Podkarpackie Center for Lung Diseases in Rzeszów,
* Patients with a history of COVID-19,
* Having obtained written informed consent (signed and dated) to participate in the study,
* Age at enrollment ≥ 18 years of age,
* No contraindications to pulmonary rehabilitation,
* No contraindications for body composition testing (bioelectrical impedance analysis).

Exclusion Criteria:

* Refusal to participate in the study,
* Patients with any acute disease in the last 3 months before baseline,
* Patients currently enrolled in any clinical trial,
* Currently infected patients with COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in the quality of life | at baseline, immediately after rehabilitation completion, and 3 months after rehabilitation completion
  Comparison of the World Health Organization Quality of Life (WHOQOL-BREF) questionnaire mean between baseline, immediately after the end of the rehabilitation protocol, and 3 months after the end of the rehabilitation protocol. The questionnaire consists of 26 questions. Answers are awarded a score in a five-point scale (1-5). Answer scores are calculated according to the WHOQOL-BREF algorithm in the range of 0-100 points. Higher score corresponds to higher quality of life.

SECONDARY OUTCOMES:
Change in lung volume parameters (spirometry) | at baseline, immediately after rehabilitation completion, and 3 months after rehabilitation completion
  Compare the results of:
  1. Forced Expiratory Volume in one second (FEV1),
  2. Forced Vital Capacity (FVC),
  3. Total Lung Capacity (TLC), and
  4. Residual volume (RV)
  between baseline, immediately after the end of rehabilitation protocol, and 3 months after the end of the rehabilitation protocol. To obtain the parameters' values, patients will perform tidal breathing and forced inspiration-expiration manoeuvre, and flow-volume loop will be recorded.
Change in respiratory flow parameters (spirometry) | at baseline, immediately after rehabilitation completion, and 3 months after rehabilitation completion
  Compare the results of:
  1. Peak Expiratory Flow (PEF) and
  2. Forced Expiratory Flow at 25-75% of vital capacity (FEF 25-75%)
  between baseline, immediately after the end of rehabilitation protocol, and 3 months after the end of the rehabilitation protocol. To obtain the parameters' values, patients will perform forced inspiration-expiration manoeuvre, and flow-volume loop will be recorded.
Change in lung diffusing capacity | at baseline, immediately after rehabilitation completion, and 3 months after rehabilitation completion
  Compare the results of Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO) [ml/min/kPa] between baseline, immediately after the end of rehabilitation protocol, and 3 months after the end of the rehabilitation protocol. To obtain parameter value, patients will perform a full inspiration of a gas mixture containing 0.3% of carbon monoxide; after ten-second breath hold patient exhales and the exhaled breath will be collected and analysed.
Change in Body Mass Index (BMI) | at baseline, immediately after rehabilitation completion, and 3 months after rehabilitation completion
  Compare the results of a BMI (kg/m^2) between baseline, immediately after the end of the rehabilitation protocol, and 3 months after the end of the rehabilitation protocol.
  To calculate BMI, the body height measurement will be performed at baseline using a stadiometer (unit: meter). Body weight will be measure at baseline, immediately after the end of the rehabilitation protocol, and 3 months after the end of the rehabilitation protocol (unit: kilogram). BMI will be calculated as body weight (kg) divided by height (m) squared.
Change in the body composition (bioelectrical impedance analysis) | at baseline, immediately after rehabilitation completion, and 3 months after rehabilitation completion
  Compare the mean content of body fat (%), fat-free mass (%), total body water (%) and muscle mass (%) between baseline, immediately after the end of the rehabilitation protocol, and 3 months after the end of the rehabilitation protocol. Body composition will be obtained using a bioelectrical impedance analysis (BIA) method by foot-to-foot body composition analyzer.
Change in C-reactive protein (CRP) values (blood sample) | at baseline, immediately after rehabilitation completion, and 3 months after rehabilitation completion
  Compare the values of C-reactive protein (CRP) [mg/dL] between baseline, immediately after the end of the rehabilitation protocol, and 3 months after the end of the rehabilitation protocol.
Change in D-Dimer values (blood sample) | at baseline, immediately after rehabilitation completion, and 3 months after rehabilitation completion
  Compare the values of D-Dimer [ng/mL] between baseline, immediately after the end of the rehabilitation protocol, and 3 months after the end of the rehabilitation protocol.
Change in white blood cell (WBC) values (blood sample) | at baseline, immediately after rehabilitation completion, and 3 months after rehabilitation completion
  Compare the values of white blood cell (WBC) [count/mm^3] between baseline, immediately after the end of the rehabilitation protocol, and 3 months after the end of the rehabilitation protocol.
Change in gasometry (blood sample) | at baseline, immediately after rehabilitation completion, and 3 months after rehabilitation completion
  Compare the values of pressures of carbon dioxide (pCO2) [mm Hg] and pressures of oxygen (pO2) [mm Hg] between baseline, immediately after the end of the rehabilitation protocol, and 3 months after the end of the rehabilitation protocol.
Change in the percentage of opacity (chest computed tomography) | at baseline, immediately after rehabilitation completion, and 3 months after rehabilitation completion
  Compare the percentage of opacity (PO%) between baseline, immediately after the end of the rehabilitation protocol, and 3 months after the end of the rehabilitation protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rzeszów / Podkarpackie Center for Lung Diseases in Rzeszów, Rzeszów, Poland